CLINICAL TRIAL: NCT02630771
Title: Multimodal Assessment of Sensory Processing and Brain Features in Patients With Chronic Orofacial Pain
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1511M80706
Record Dates: First submitted 2015-12-02; First posted 2015-12-15 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Toothache; Temporomandibular Joint Disorders
MeSH Terms: conditions — Toothache; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PDAP only: Persistent dentoalveolar pain disorder patients who do not fit criteria for TMD. Pressure pain threshold before/during conditioned pain modulation.
  Interventions: Procedure: Pressure pain threshold
- PDAP + TMD: Persistent dentoalveolar pain disorder patients who also fit criteria for TMD. Pressure pain threshold before/during conditioned pain modulation.
  Interventions: Procedure: Pressure pain threshold
- Painfree controls: Painfree subjects. Pressure pain threshold before/during conditioned pain modulation.
  Interventions: Procedure: Pressure pain threshold

INTERVENTIONS:
Procedure: Pressure pain threshold — Pressure algometry over thenar eminence, bilateral masseter muscles measured at baseline and during conditioned pain modulation
  Other Names: PPT

SUMMARY:
This proposal will investigate pain modulatory mechanisms and brain functional and structural characteristics using multiple MRI modalities in persistent dentoalveolar pain disorder (PDAP) patients with and without temporomandibular disorders (TMD). All measures from patients will be compared to painfree controls.

DETAILED DESCRIPTION:
Chronic orofacial pain disorders may present localized in the mouth such as with persistent dentoalveolar pain disorder (PDAP) or widespread in the head/face/jaw such as with temporomandibular disorders (TMD). PDAP pain manifests in a tooth that usually underwent root canal treatment or in the site formally occupied by such tooth, while TMD pain is usually reported over the preauricular area, jaws and temples. These commonly comorbid disorders have a significant impact on the individual and society. Their mechanisms are poorly understood with evidence suggesting deficient pain modulation and abnormal brain features. PDAP and TMD patients, when compared to controls, have abnormal sensory/pain processing as well as brain structural and functional differences.

This proposal will investigate pain modulatory mechanisms and brain functional and structural characteristics using multiple MRI modalities in PDAP patients with and without TMD. All measures from patients will be compared to painfree controls. This knowledge will support better understanding of mechanisms involved in PDAP and will support development of mechanistic-based clinical treatments for the patients the investigators serve. Findings from these investigations will likely contribute to our understanding of other chronic pain conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age- and handedness-matched painfree controls using frequency matching to maintain similar group averages:

   * No self-report of persistent pain conditions for the last 6 months;
   * No diagnosis of PDAP or TMD;
2. PDAP only:

   * Fulfilling diagnostic criteria per Nixdorf et al., 20122
   * Characteristic dentoalveolar PDAP pain cannot be increased by pressure provocation from jaw muscle trigger points (referred pain)
3. PDAP with TMD:

   * Fulfilling diagnostic criteria for PDAP2 and chronic TMD myalgia per Schiffman et al. 20143

Exclusion Criteria:

Self-report:

1. Chronic widespread pain
2. Current use of opioids or other pain medications (e.g., ibuprofen/acetaminophen) that cannot be stopped <3 days prior to testing
3. Conditions/diseases associated with altered pain perception: neurological (e.g., multiple sclerosis, trigeminal neuralgia) psychiatric disorders, diabetes, neoplasm and cardiovascular disorders
4. Injury to hands
5. Substance abuse
6. MRI contraindications including pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Females with age range 18-65 years
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-01; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold change before and during conditioned pain modulation | Baseline
  Pressure pain thresholds will be determined over the skin overlaying the masseter muscles bilaterally and over the right thenar eminence using a pressure algometer before and during the application of a concurrent noxious heat stimulus to the left forearm.

CONTACTS AND LOCATIONS:
Overall Officials: Estephan J Moana-Filho, DDS, MS, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota School of Dentistry, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided